CLINICAL TRIAL: NCT06424418
Title: A Proof of Concept Study Validating The Safety And Efficacy of a Novel Robotic Scope Cleaner
Brief Title: Robotic Scope Cleaning Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boehringer Labs LLC (Industry)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Scope1
Record Dates: First submitted 2024-04-26; First posted 2024-05-22 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Robotic Scope Cleaner — The device is used to clean the scope when it visualization becomes obstructed during a surgical procedure.

SUMMARY:
A novel device that works with robotic trocars to clean the scope when visualization is compromised during a surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* able to consent
* undergoing a surgical robotic procedure

Exclusion Criteria:

* not suitable for a surgical procedure with the robot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
feasibility of device | [Estimated 6 months]
  Study to determine if the device works as intended. A questionnaire will be filled out by the operating surgeon. Questions include the number of cleans, time to clean, ease of use, etc.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No